CLINICAL TRIAL: NCT06342076
Title: Comparison of the Efficacy of Subcostal Transversus Abdominis Plane Block and Rectus Sheath Block for Postoperative Analgesia in Major Open Gynaecological Cancer Surgery: a Prospective Randomised Study
Brief Title: Comparison of the Efficacy of Peripheral Nerve Blocks in Major Open Gynaecological Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-596
Record Dates: First submitted 2024-03-21; First posted 2024-04-02 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pain; Postoperative Complications; Analgesia; Regional Anesthesia Morbidity
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Agnosia

STUDY DESIGN:
Intervention Model Description: Prospective randomize study
Masking Description: Prospective randomize study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1: Subcostal transversus abdominis plane block(STAPB) (Experimental): Subcostal transversus abdominis plane block(STAPB)
  Interventions: Procedure: Patients undergoing subcostal transversus abdominis plane block and posterior transversus abdominis plane block; Procedure: Patients undergoing rectus sheat block and posterior transversus abdominis plane block
- Group 2: Rectus sheat block(RSB) (Experimental): Rectus sheat block(RSB)
  Interventions: Procedure: Patients undergoing subcostal transversus abdominis plane block and posterior transversus abdominis plane block; Procedure: Patients undergoing rectus sheat block and posterior transversus abdominis plane block

INTERVENTIONS:
Procedure: Patients undergoing subcostal transversus abdominis plane block and posterior transversus abdominis plane block — To prevent postoperative pain, the researchers applied a subcostal transversus abdominis plane block in addition to the posterior transversus abdominis plane block to a group of patients who underwent surgery with a midline incision due to major gynecological cancer.
Procedure: Patients undergoing rectus sheat block and posterior transversus abdominis plane block — To prevent postoperative pain, the researchers applied a rectus sheath block in addition to the posterior transversus abdominis plane block to a group of patients who were operated on through a midline incision due to major gynecological cancer.

SUMMARY:
The aim of this prospective randomized study was to compare the effectiveness of subcostal transversus abdominis plane block or rectus sheath block applied in addition to posterior transversus abdominis plane block for postoperative analgesia in major gynecological cancer surgeries.

The main question(s) it aims to answer are:

[Is subcostal transversus abdominis plane block more effective in postoperative analgesia? ] [Is there a difference in pain scores at 24 hours after surgery? ] Since pain scores within the first 24 hours after surgery will be evaluated, participants will be asked to give a value between 0 and 10 at certain time periods.

DETAILED DESCRIPTION:
This prospective, randomized study was conducted at Başakşehir Çam and Sakura City Hospital in accordance with the Declaration of Helsinki. After ethics committee approval (decision no: 2023-596, date: 22.11.2023) and written consent from all patients, the study was conducted according to Consolidated Standards of Reporting Trials (CONSORT) guidelines. In the study, which included a total of 50 patients, the patients were divided into two groups: subcostal transversus abdominis plane block (STAPB) or rectus sheath block (RSB). Postoperative 24-hour VAS values, opioid demand and administration amounts in intravenous patient-controlled analgesia, presence of nausea and vomiting, surgical complications and length of hospital stay were evaluated (6th hour, 12th hour, 24th hour).

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* ASA II-III

Exclusion Criteria:

* Those who are allergic to local anesthetics
* BMI> 40 kg/m2
* Those with chronic pain
* Those with a history of previous abdominal surgery
* Patients who refuse the use of postoperative patient-controlled analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
visuel analog scale | 24 hours postoperatively
  Our primer aim was to compare postoperative pain scores. The first 24 hours postoperatively were evaluated.Numeric Rating Scale(NRS) was used to assess postoperative pain.6th, 12th, 24th hour NRS values were recorded For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
amount of opioid used | 24 hours postoperatively
  Our secondary aim was to evaluate the opioid amount (mg) in the first 24 hours of intravenously administered opioids with patient-controlled analgesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Basaksehir, Turkey (Türkiye)

REFERENCES:
- [Result] Bhatia N, Arora S, Jyotsna W, Kaur G. Comparison of posterior and subcostal approaches to ultrasound-guided transverse abdominis plane block for postoperative analgesia in laparoscopic cholecystectomy. J Clin Anesth. 2014 Jun;26(4):294-9. doi: 10.1016/j.jclinane.2013.11.023. Epub 2014 Jun 2. PMID 24882606
- [Result] Hebbard PD, Barrington MJ, Vasey C. Ultrasound-guided continuous oblique subcostal transversus abdominis plane blockade: description of anatomy and clinical technique. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):436-41. doi: 10.1097/aap.0b013e3181e66702. PMID 20830871
- [Result] Yorukoglu HU, Sahin T, Oge Kula A. Transversus Abdominis Plane Block Versus Rectus Sheath Block for Postoperative Pain After Caesarean Delivery: A Randomised Controlled Trial. Turk J Anaesthesiol Reanim. 2023 Feb;51(1):43-48. doi: 10.5152/TJAR.2023.22724. PMID 36847318
- [Result] Soliz JM, Lipski I, Hancher-Hodges S, Speer BB, Popat K. Subcostal Transverse Abdominis Plane Block for Acute Pain Management: A Review. Anesth Pain Med. 2017 Oct 20;7(5):e12923. doi: 10.5812/aapm.12923. eCollection 2017 Oct. PMID 29696110
- [Result] Abdelsalam K, Mohamdin OW. Ultrasound-guided rectus sheath and transversus abdominis plane blocks for perioperative analgesia in upper abdominal surgery: A randomized controlled study. Saudi J Anaesth. 2016 Jan-Mar;10(1):25-8. doi: 10.4103/1658-354X.169470. PMID 26955306